CLINICAL TRIAL: NCT03260478
Title: HEMOglobin Transfusion Threshold in Traumatic Brain Injury OptimizatioN: The HEMOTION Trial
Acronym: HEMOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Critical Care Trials Group (Other); Canadian Traumatic Brain Injury Research Consortium (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Perioperative Anesthesia Clinical Trials (PACT) Group (Unknown)
Responsible Party: Principal Investigator, Dr Alexis Turgeon, Professor, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-20-2018-3706
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury; Transfusion
Keywords: Traumatic Brain Injury (TBI); Red Blood Cells (RBC) Transfusion; Intensive Care Unit (ICU); Transfusion Threshold; Anemia; Oxygen Delivery; Neurocritical Care; Critical Care Neurology and Trauma
MeSH Terms: conditions — Brain Injuries, Traumatic; Anemia; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-label with blinded outcome evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal Transfusion Strategy (Experimental): Patients will receive red blood cells transfusion if Hb ≤ 100 g/L.
  Interventions: Procedure: Red Blood Cells Transfusion
- Restrictive Transfusion Strategy (Experimental): Patients will receive red blood cells transfusion if Hb ≤ 70 g/L.
  Interventions: Procedure: Red Blood Cells Transfusion

INTERVENTIONS:
Procedure: Red Blood Cells Transfusion — Transfusion of packed red blood cells unit(s).

SUMMARY:
Most trauma deaths are related to traumatic brain injury (TBI). Although the management of patients has improved, mortality remains unacceptably high, and half of survivors of moderate and severe TBI are left with major functional impairment. Current management guidelines are based on limited evidence and practice is highly variable. Most acutely ill patients with TBI will develop anemia, which may decrease oxygen delivery to a fragile brain. While clinical practice is moving towards transfusing at low hemoglobin (Hb) levels, experts have expressed concerns regarding restrictive strategies, which may adversely affect clinical outcomes in TBI. Our primary objective is to evaluate the effect of red blood cell (RBC) transfusion thresholds on neurological functional outcome. We hypothesize that a liberal transfusion strategy improves outcomes compared to a restrictive strategy.

ELIGIBILITY:
Inclusion Criteria:

* Acute moderate to severe blunt TBI
* Glasgow Coma Score [GCS] ≤ 12
* Hb level ≤ 100 g/L

Exclusion Criteria:

* Patient has received transfusion after ICU admission
* Contraindications or known objection to transfusions
* Glasgow Coma Scale (GCS) of 3 with dilated fixed pupils.
* Patient is brain dead
* Active life-threatening bleeding with hemorrhagic shock or requiring urgent surgical procedure
* A decision to withold or withdraw life-sustaining therapies was made
* No fixed address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
extended Glasgow Outcome Scale (GOSe) | 6 months
  Assessment of neurological outcome by the extended Glasgow Outcome Scale (GOSe)

SECONDARY OUTCOMES:
Mortality | ICU, Hospital and at 6 months
  Assessment of patient mortality.
Functional Independence Measure (FIM) | 6 months
  Assessment of patient function.
Quality of life (EQ-5D) | 6 months
  Evaluation of the overall quality of life.
Quality of life (Qolibri questionnaires) | 6 months
  Evaluation of the quality of life specific to the TBI.
Depression (PHQ-9) | 6 months
  Assessment of depression.

OTHER OUTCOMES:
Number RBC transfusions | While in the ICU, censored at 6 months after randomization
  Assessment of the number of RBC transfusions.
Lowest Daily Hemoglobin | While in the ICU, censored at 6 months after randomization
  Assessment of the Median Lower Daily Hemoglobin.
Infections | While in the ICU, censored at 6 months after randomization
  Assessment of the incidence of infections.
Duration of mechanical ventilation | While in the ICU, censored at 6 months after randomization
  Duration of mechanical ventilation.
ICU Lenght of stay | While in the ICU, censored at 6 months after randomization
  Lenght of stay in the intensive care unit
Hospital Lenght of stay | While in the hospital, censored at 6 months after randomization
  Duration of hospitalization is study hospital
Complications related to transfusion | While in the ICU, censored at 6 months after randomization
  Assessment of complications related to RBC transfusions.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Turgeon, MD MSc FRCPC, Principal Investigator — CHU de Quebec-Université Laval Research Center; François Lauzier, MD MSc FRCPC, Principal Investigator — CHU de Quebec-Université Laval Research Center; Dean Fergusson, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (33):
- Brazil (2):
  - Santa Casa de Misericórdia de Barretos, Barretos, São Paulo
  - The Hospital das Clinicas da Facudade de Medicina da USP, São Paulo
- Canada (18):
  - Foothills Medical Center, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Winnipeg Health Sciences Center, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Center, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Center, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - CIUSSS De l'Estrie, Sherbrooke, Quebec
  - CIUSSS Mauricie-et-Centre-du-Québec, Trois-Rivières, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - CHU de Québec-Université Laval (Hôpital de l'Enfant-Jésus), Université Laval, Québec
- France (4):
  - CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - CHU de Besançon, Besançon, Bourgogne-Franche-Comté
  - Hôpital de Hautepierre, Strasbourg, Grand Est
  - CHU de Nîmes, Nîmes, Occitanie
- United Kingdom (9):
  - University Hospital of Wales, Cardiff
  - Western General Hospital, Edinburgh
  - Aintree University Hospital, Liverpool
  - Walton Centre, Liverpool
  - St. Mary's Hospital (Imperial College Healthcare), London
  - James Cook University Hospital, Middlesbrough
  - University of Nottingham Hospital, Nottingham
  - Salford Royal Hospital, Salford
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Turgeon AF, Fergusson DA, Clayton L, Patton MP, Neveu X, Walsh TS, Docherty A, Malbouisson LM, Pili-Floury S, English SW, Zarychanski R, Moore L, Bonaventure PL, Laroche V, Verret M, Scales DC, Adhikari NKJ, Greenbaum J, Kramer A, Rey VG, Ball I, Khwaja K, Wise M, Harvey D, Lamontagne F, Chabanne R, Algird A, Krueper S, Pottecher J, Zeiler F, Rhodes J, Rigamonti A, Burns KEA, Marshall J, Griesdale DE, Sisconetto LS, Kutsogiannis DJ, Roger C, Green R, Boyd JG, Wright J, Charbonney E, Nair P, Astles T, Sy E, Hebert PC, Chasse M, Gomez A, Ramsay T, Taljaard M, Fox-Robichaud A, Tinmouth A, St-Onge M, Costerousse O, Lauzier F; HEMOTION Trial Investigators on behalf of the Canadian Critical Care Trials Group, the Canadian Perioperative Anesthesia Clinical Trials Group, and the Canadian Traumatic Brain Injury Research Consortium. Liberal or Restrictive Transfusion Strategy in Patients with Traumatic Brain Injury. N Engl J Med. 2024 Aug 22;391(8):722-735. doi: 10.1056/NEJMoa2404360. Epub 2024 Jun 13. PMID 38869931
- [Derived] Turgeon AF, Fergusson DA, Clayton L, Patton MP, Zarychanski R, English S, Docherty A, Walsh T, Griesdale D, Kramer AH, Scales D, Burns KEA, Boyd JG, Marshall JC, Kutsogiannis DJ, Ball I, Hebert PC, Lamontagne F, Costerousse O, St-Onge M, Lessard Bonaventure P, Moore L, Neveu X, Rigamonti A, Khwaja K, Green RS, Laroche V, Fox-Robichaud A, Lauzier F; HEMOTION Trial Team, the Canadian Critical Care Trials Group, the Canadian Perioperative Anesthesia Clinical Trials Group and the Canadian Traumatic Brain Injury Research Consortium. Haemoglobin transfusion threshold in traumatic brain injury optimisation (HEMOTION): a multicentre, randomised, clinical trial protocol. BMJ Open. 2022 Oct 10;12(10):e067117. doi: 10.1136/bmjopen-2022-067117. PMID 36216432
- See also: Canadian Traumatic Brain Injury Research Consortium website — https://www.ctrc-ccrt.ca
- Available data/document: Study Protocol — https://bmjopen.bmj.com/content/12/10/e067117.info

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03260478/SAP_001.pdf